CLINICAL TRIAL: NCT00913367
Title: A Multi-center, Open, Randomized, Parallel-group, 2 Arm Study to Compare the Efficacy and Safety of Amaryl®M 1/500mg Twice Daily Versus Amaryl® 4mg Both in Combination With Lantus® Once-daily Regimen in Type 2 Diabetes Mellitus Patients With Inadequate Glycemic Control
Brief Title: Efficacy/Safety Study of Amaryl®M 1/500 mg Twice Daily Versus Amaryl® 4 mg Both in Combination With Lantus® in Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Handok Inc. (Industry)
Responsible Party: Moon Hwa Park / Medical Research Team Manager, Medical Research Team
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HANDOK2008.10
Record Dates: First submitted 2009-05-26; First posted 2009-06-04 (Estimated); Last update posted 2013-03-28 (Estimated); Status verified 2013-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — glimepiride; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amaryl group (Active Comparator)
  Interventions: Drug: glimepiride + insulin glargine (Amaryl + Lantus)
- Amaryl M group (Experimental)
  Interventions: Drug: glimepiride/metformin fixed combination+insulin glargine (AmarylM + Lantus)

INTERVENTIONS:
Drug: glimepiride + insulin glargine (Amaryl + Lantus) — * Amaryl® 4 mg at breakfast + Lantus® at dinner
  * The initial dose of Lantus® is 0.2IU/kg at baseline. Lantus® titration will be made by patients every 3 days based on the mean value of previous 3 fasting SMBG level before breakfast
  Other Names: Amaryl; Lantus injection solostar
  Arms: Amaryl group
Drug: glimepiride/metformin fixed combination+insulin glargine (AmarylM + Lantus) — * Amaryl® M 1/500 mg at breakfast + Amaryl® M 1/500 mg at dinner + Lantus® at dinner
  * The initial dose of Lantus® is 0.2IU/kg at baseline. Lantus® titration will be made by patients every 3 days based on the mean value of previous 3 fasting SMBG level before breakfast
  Other Names: Amaryl M; Lantus injection solostar
  Arms: Amaryl M group

SUMMARY:
The purpose of this study is to compare the efficacy of Amaryl®M 1/500 mg twice daily versus Amaryl® 4 mg both in combination with Lantus® once-daily regimen in type 2 Diabetes Mellitus patients with inadequate glycemic control.

DETAILED DESCRIPTION:
There are several kinds of oral antidiabetic drugs (OADs) that are used in the treatment of patients with type 2 DM. Among them, sulfonylurea and metformin are well-established first-line OADs. However, as the beta cell dysfunction progresses over time, patients fail to achieve good glycemic control with OADs alone and need further treatment intensification, usually involving the introduction of insulin either alone or in combination with OADs. Now, an OAD combined with bedtime insulin is one of the recommended treatment options for patients with type 2 DM and OAD failure. But, it still remains unclear which OADs are the most effective in combination with insulin for the treatment of type 2 DM.

so, this study we will be able to verify which OADs are the most effective in combination with insulin for the treatment of type 2 DM.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 20 years old with type 2 DM
* Patients with inadequate glycemic control despite continuous use of tolerable or maximal doses of one or more OADs for 3months or more.
* 7%<HbA1c<11 % at screening
* 21 kg/m2 ≤ BMI ≤ 30 kg/m2
* Patents who need insulin add-on therapy based on investigator's discretion
* Patients who would give the informed consent
* Patients who can perform SMBG and record the data on the patient's diary

Exclusion Criteria:

* History of acute metabolic complications such as diabetic ketoacidosis or hyperosmolar nonketotic coma within 3 months before screening
* Pregnant or lactating females
* History of drug or alcohol abuse
* Patients with known hypersensitivity to glimepiride, metformin HCL or insulin
* Night-shift workers
* Patients who are under insulin therapy at screening
* Treatment with any investigational products in the last 3 months before screening
* Clinically significant laboratory abnormality on screening labs or any medical condition that would affect the completion or outcome of the study based on investigator's decision
* Patients with serum creatinine level > 1.5 mg/dl in male and > 1.4 mg/dl in female
* Patients with ALT or AST > 3x ULN

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Mean change in HbA1c from baseline to the last visit | 16 weeks

SECONDARY OUTCOMES:
Mean change in FPG, insulin, c-peptide from baseline to the last visit Safety; Episodes of hypoglycemia & other adverse events | 16 weeks
Response rate based on HbA1c and FPG levels measured at the last visit | 16 weeks
Mean change in Lantus® dose from baseline to the last visit | 16 weeks
Compliance | 16 weeks
Frequency with hypoglycemic episode | 16weeks
Adverse events | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kang S Park, Principal Investigator — Eulji University Hospital
Locations (1):
- HeeYoung Lee, Seoul, South Korea